CLINICAL TRIAL: NCT01601431
Title: The Utility of Cap Colonoscopy in Increasing Adenoma Detection Rate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was inactivated by the IRB since PI left institution.
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Mohamed O Othman, Principal Investigator, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E12050
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Adenoma
Keywords: Screening colonoscopy
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cap Assisted Colonoscopy (Experimental): Cap Assisted Colonoscopy uses a Cap which is a transparent hood which is attached to the distal end of the colonscope and allows depressing the colon folds in order to visualize hidden polyps behind the folds.
  Interventions: Device: Cap Assisted Colonoscopy
- Conventional colonoscopy (Active Comparator): A conventional colonoscopy does not use a Cap in order to perform the procedure
  Interventions: Device: Conventional colonoscopy

INTERVENTIONS:
Device: Cap Assisted Colonoscopy — Plastic transparent cap added to the distal end of the colonoscope which can increase adenoma detection rate
  Arms: Cap Assisted Colonoscopy
Device: Conventional colonoscopy — Regular colonoscopy as per standard clinical guidelines
  Arms: Conventional colonoscopy

SUMMARY:
This is a research study about the usefulness of transparent cap during screening colonoscopy. The purpose of the research is to test the usefulness of adding small cap to the tip of the colonoscope. the investigators hypothesis is that Cap assisted colonoscopy will improve the detection of adenomatous polyps (polyps which can become colon cancer later on) in comparison to the standard colonoscopy.

DETAILED DESCRIPTION:
This is a prospective, randomized trial comparing the adenoma detection rate between Hispanic patients undergoing a screening colonoscopy with a conventional colonoscope or with a cap-assisted colonoscopy. The aims of the study are:

1. Compare ADR between Hispanic patients undergoing a screening colonoscopy with and without cap.
2. Compare the overall polyp detection rate between Hispanic patients undergoing a screening colonoscopy with and without cap.
3. Compare the cecal intubation rate and cecal intubation time between standard colonoscopy and cap assisted colonoscopy.
4. Compare the complication rate between standard colonoscopy and cap assisted colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Hispanic patients (18-80) who are undergoing colonoscopy for screening or surveillance purposes.

Exclusion Criteria:

1. Patients younger than 18 yrs old or older than 80 yrs.
2. Patients with a prior history of colonic surgeries
3. Patient with Crohns colitis or ulcerative colitis.
4. Patient with prior history of colon cancer
5. Patient with poor bowel preparation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2012-03-29 (Actual); Primary Completion 2015-02-02 (Actual); Study Completion 2015-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed O Othman, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cap Assisted Colonoscopy | Conventional Colonoscopy
Started | 223 | 217
Completed | 211 | 214
Not Completed | 12 | 3

BASELINE CHARACTERISTICS:
Groups:
- Conventional Colonoscopy: A conventional colonoscopy does not use a Cap in order to perform the procedure
  Cap Assisted Colonoscopy: Plastic transparent cap added to the distal end of the colonoscope which can increase adenoma detection rate
  Conventional colonoscopy: Regular colonoscopy as per standard clinical guidelines
- Total: Total of all reporting groups
Arm/Group | Cap Assisted Colonoscopy | Conventional Colonoscopy | Total
Number analyzed (Participants) | 223 | 217 | 440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 220 | 212 | 432
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.48 (7.28) | 60.08 (7.26) | 60 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 155 | 301
  Male | 77 | 62 | 139
Adenoma Detection Rate [Count of Participants; unit: Participants] | 66 | 69 | 135
Polyp detection rate [Count of Participants; unit: Participants] | 87 | 92 | 179
Advanced adenoma detection rate [Count of Participants; unit: Participants] | 21 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: ADR Differences in Hispanic Patients Undergoing a Screening Colonoscopy With and Without Cap.
Description: 1. Compare ADR between Hispanic patients undergoing a screening colonoscopy with and without cap.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cap Assisted Colonoscopy | Conventional Colonoscopy
Number analyzed (Participants) | 211 | 214
Participants | 66 | 69

ADVERSE EVENTS:
Arm/Group | Cap Assisted Colonoscopy | Conventional Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/214
Serious Adverse Events (participants affected / at risk) | 1/211 | 0/214
Other Adverse Events (participants affected / at risk) | 0/211 | 0/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cap Assisted Colonoscopy (N=211) | Conventional Colonoscopy (N=214)
Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
single center study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes